CLINICAL TRIAL: NCT05845307
Title: Randomized Pre-surgical Window-of-Opportunity Trial of TTI-101 in Patients With Stage II-IV Resectable HPV-negative Squamous Cell Carcinoma of the Head and Neck
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: 0 participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Tvardi Therapeutics, Inc (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0001; NCI-2023-03573 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Control Groups; C188-9 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Experimental): Participants you will be randomly assigned to either receive the study drug or be in a control group.
  Interventions: Drug: Control Group
- TTI-101 (Experimental): Participants you will be randomly assigned to either receive the study drug or be in a control group.
  Interventions: Drug: TTI-101

INTERVENTIONS:
Drug: Control Group — Given by PO
  Arms: Control Group
Drug: TTI-101 — Given by PO
  Arms: TTI-101

SUMMARY:
To learn if TTI-101 can reduce the growth of HPV-negative squamous cell carcinomas of the head and neck when given before standard of care surgery.

DETAILED DESCRIPTION:
Objectives:

Primary:

• To determine the change in pY-STAT3 H-score in tumor tissue in post-treatment resection specimens versus pre-treatment biopsy specimens.

Secondary:

* To determine the safety and tolerability of pre-surgery TTI-101 in patients with Stage II-IV HPV-negative HNSCC who are planned for definitive local surgery with or without radiation.
* To determine the individual pre/post treatment changes in pY-STAT3 H-scores in epithelial and stromal tumor cells.
* To determine the pathologic response rate to pre-surgery TTI-101.
* To determine the overall response rate (ORR) to pre-surgery TTI-101 using RECIST v1.1 criteria.
* To determine the disease free, disease specific and overall survival (DFS, DSS, OS) after pre-surgery TTI-101 treatment and SOC surgery.

Exploratory:

* To evaluate the effects of pre-surgery TTI-101 on circulating and tumor-infiltrating immunocytes, and on the intratumoral expression of PD-1 along with other immune related molecules.
* To compare outcome measures (response rate and survival) in control versus TTI-101-treated patients.
* To determine the association of immunologic changes with treatment response.
* To determine the association of pharmacokinetic (PK) measures with treatment response.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Biopsy-proven primary Stage II-IV squamous cell carcinoma of the head and neck
* For oropharyngeal cancer patients: HPV-negative by p16 and/or direct high-risk HPV assessment
* Surgical resection must be planned as primary therapy with or without adjuvant radiation therapy.
* Signed Informed Consent Form (ICF).
* Ability and willingness to comply with the requirements of the study protocol.
* Ability to swallow study drug.
* Age years of 18 years.
* Measurable disease per RECIST v1.1 (see Appendix 2) and/or per direct clinical measurements.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (see Appendix 4)
* Adequate hematologic and hepatorenal function, defined by the following laboratory results obtained within 4 weeks prior to study entry:

  * ANC 1500 cells/L
  * Platelet count 100,000/L;
  * Hemoglobin 9.0 g/dL
  * Total bilirubin 1.5 upper limit of normal (ULN) with the following exception:

Patients with known Gilbert disease who have serum bilirubin level 3 ULN may be enrolled.

* AST and ALT 2.5 ULN
* Alkaline phosphatase 2.5 ULN
* Serum creatinine clearance ≥60 mL/min, measured or calculated per institutional standard protocol

  • INR and aPTT 1.5 ULN
* This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.

  * No evidence of distant metastases.
  * A male participant must agree to use contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.
  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
  * Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
  * A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 90 days after the last dose of study treatment.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry.

General Exclusion Criteria:

* Any prior systemic or radiotherapy within the last 4 months directed towards the squamous cell carcinoma of the head and neck that is to be resected as part of SOC therapy.
* Standard of care anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, for concurrent malignancy or unresected squamous cell carcinoma of the head and neck within 3 weeks prior to initiation of study treatment.
* AEs from prior anticancer therapy that have not resolved to Grade 1 except for alopecia, Grade 2 neuropathy or endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement are eligible
* Pregnancy, lactation, or breastfeeding
* Inability to comply with study and follow-up procedures
* Has a known active Hepatitis B (defined as Hepatitis B RNA detected) or known active Hepatitis C virus (defined as HCV RNA is detected) infection, or known active HIV (defined as HIV RNA is detected) infection.
* Active tuberculosis
* Severe infections within 4 weeks prior to treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection as determined by the treating team within 2 weeks prior to treatment
* Major surgical procedure within 28 days prior to treatment
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed or mRNA vaccines is allowed.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, well-differentiated thyroid cancer, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
* History of significantly impaired cardiac function such as unstable angina pectoris, congestive heart failure with New York Heart Association (NYHA) class III or IV, myocardial infarction within the last 12 months prior to trial entry; signs of pericardial effusion, serious arrhythmia (including QTc prolongation of >470 ms and/or pacemaker) or prior diagnosis of congenital long QT syndrome or left ventricular ejection fraction <50% on echocardiogram.
* History of cerebral vascular accident or stroke within the previous 2 years.
* Uncontrolled hypertension (>160/100mm Hg).
* History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemicalor biologic composition as TTI-101 (hydroxyl-naphthalene sulfonamides).
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Previous treatment of the current malignancy with a STAT inhibitor.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Medication-Related Exclusion Criteria:

* Bisphosphonate therapy for symptomatic hypercalcemia

  - Use of bisphosphonate therapy for other reasons (e.g., osteoporosis) is allowed.
* Received oral or IV antibiotics within 2 weeks prior to treatment

  - Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Treatment with an investigational agent (not standard of care) within 3 weeks prior to treatment (or within five halflives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to treatment

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sikora, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT05845307/ICF_000.pdf